CLINICAL TRIAL: NCT02123550
Title: Doppler Ultrasound Imaging of Plastic Surgery Patients for Deep Venous Thrombosis Detection: A Prospective Controlled Study.
Brief Title: Doppler Ultrasound Imaging of Plastic Surgery Patients for DVT Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swanson Center (Other)
Responsible Party: Sponsor
Other Study IDs: Swanson01
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Deep Venous Thrombosis
Keywords: deep; venous; thrombosis; Doppler; ultrasound; plastic; surgery; thromboembolism; prevention
MeSH Terms: conditions — Venous Thrombosis; Thrombosis; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective controlled study examines the use of Doppler ultrasound as a means to screen elective plastic surgery patients for the presence of deep venous blood clots both before and after surgery. This is a noninvasive technique that is known to be both sensitive and specific for the detection of deep venous thromboses in the lower extremities. This method may make it unnecessary to select patients for prophylactic anticoagulation, which poses additional risks to the patient.

DETAILED DESCRIPTION:
Protocol

Investigation of Deep Venous Thromboses in Elective Cosmetic Surgery Patients using Doppler Ultrasound

Background/Purpose

Venous thromboembolism is a well-known and serious risk of surgery. In an attempt to reduce the frequency of this postoperative complication, many plastic surgeons today elect to anticoagulate patients deemed to be at higher risk.1 The efficacy and ethics of this treatment have been challenged.2 Moreover, prophylactic anticoagulation poses additional serious risks of its own, including increased bleeding and wound hematomas.2 It makes sense to use a screening device to detect not just symptomatic cases but also subclinical deep venous thrombosis so that treatment can be promptly initiated and patients without evidence of blood clots can be spared the needless side effects of anticoagulation.

Doppler ultrasound imaging represents a sensitive, direct, and noninvasive method to screen for the presence of venous thromboses.3 This prospective study is undertaken to determine its feasibility in the setting of outpatient plastic surgery. Doppler ultrasound imaging as a screening tool for elective plastic surgery patients has not been previously published. This test is added to the perioperative protocol, which is otherwise unchanged.

Subjects

Two hundred consecutive consenting adult men and women undergoing outpatient elective plastic surgery under total intravenous anesthesia will be investigated using Doppler ultrasound scans preoperatively, on the first day after surgery, and approximately 1 week after surgery. Common operations included liposuction, abdominoplasty, facelifts, and cosmetic breast surgery. In addition, 25 control patients (i.e., men and women not having surgery) will be investigated at the same intervals.

Scans

The Terason t3200 Ultrasound System Vascular series images the deep veins of both lower extremities. The veins evaluated with this imaging technique consist of the common femoral, greater saphenous, superficial femoral, popliteal, and posterior tibial veins. Both color Doppler flow and 2-dimensional compression tests (Duplex scans) are performed. The thickness of the adipose layer is also measured and patient weights are recorded to check for any possible correlations.

Clinical measures to reduce the risk of venous thrombosis include: (1) spontaneous breathing without muscle relaxants, (2) no prone positioning in surgery, (4) sequential compression devices, (4) movement of the lower extremities during surgery, and (5) outpatient treatment with early ambulation.2

Patients are cautioned that deep venous thrombosis (blood clots) are a known risk of surgery and that they are to report any asymmetrical swelling of the lower extremities, thigh pain, or fever to their surgeon immediately. Any patient with a positive scan is referred to a local hospital for confirmation and treatment.

Null Hypothesis

Ultrasound scans are a safe, noninvasive, effective method to detect blood clots in the deep veins of the lower extremities in plastic surgical patients.

Informed Consent

Patients are informed as to the nature of the study and are told that their participation is entirely voluntary and they are free to decline, and that doing so does not in any way prejudice their treatment.

Patient Risk

There is no patient risk. The study does not affect patient treatment. It offers the possibility of detection of sub-clinical deep venous thrombosis.

Sample Size

A sample of 2000 treated patients and 25 controls is anticipated.

Disclosure

The author has no financial interest in any of the products, devices, or drugs mentioned in this article. The author has no conflicts of interest to disclose. There was no outside funding for this study.

ELIGIBILITY:
Inclusion Criteria:

* elective plastic surgery patient
* consenting patient

Exclusion Criteria:

* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2000 study patients consisting of consecutive elective patients undergoing outpatient plastic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01; Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Sonographic evidence of a thrombosis | 1 week
  Doppler ultrasound is used to detect evidence of a deep venous thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Swanson, M.D., Principal Investigator — Swanson Center
Locations (1):
- Swanson Center, Leawood, Kansas, United States

REFERENCES:
- [Background] Pannucci CJ, Dreszer G, Wachtman CF, Bailey SH, Portschy PR, Hamill JB, Hume KM, Hoxworth RE, Rubin JP, Kalliainen LK, Pusic AL, Wilkins EG. Postoperative enoxaparin prevents symptomatic venous thromboembolism in high-risk plastic surgery patients. Plast Reconstr Surg. 2011 Nov;128(5):1093-1103. doi: 10.1097/PRS.0b013e31822b6817. PMID 22030491
- [Derived] Swanson E. Prospective Study of Doppler Ultrasound Surveillance for Deep Venous Thromboses in 1000 Plastic Surgery Outpatients. Plast Reconstr Surg. 2020 Jan;145(1):85-96. doi: 10.1097/PRS.0000000000006343. PMID 31881608